CLINICAL TRIAL: NCT04251429
Title: Safety and Health Through Integrated Facilitated Teams (SHIFT)
Brief Title: Effectiveness of the Healthy Workplace Participatory Program with Peer-led Teams in Public Sector Healthcare Facilities
Acronym: SHIFT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alicia Kurowski, Research Professor, University of Massachusetts, Lowell
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: U19OH008857 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2020-01-31 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Work-Related Condition; Burnout, Caregiver; Work-related Injury; Musculoskeletal Pain
Keywords: participatory; employee engagement; process evaluation; work ability
MeSH Terms: conditions — Caregiver Burden; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention Group (Experimental): SHIFT study team provides coaching to Health and Safety Committee to implement a participatory program for increasing committee effectiveness.
  Interventions: Other: CPH-NEW Healthy Workplace Participatory Program
- Delayed Intervention Group (Other): Active Comparator for 2 years: status quo program remains in place with new ongoing data collection. Then experimental intervention as above.
  Interventions: Other: CPH-NEW Healthy Workplace Participatory Program

INTERVENTIONS:
Other: CPH-NEW Healthy Workplace Participatory Program — A participatory program for increasing effectiveness of occupational health and safety committees or peer-led employee teams through root cause analysis, prioritizing health and safety needs for effective problem-solving, identifying feasible interventions, and presenting these to senior leadership. Interventions are selected and implemented by leadership and evaluated by both teams.

SUMMARY:
Safety & Health through Integrated, Facilitated Teams (SHIFT) is an intervention study to enhance employee health, safety, and well-being in public sector healthcare institutions in New England. The investigators will evaluate the effectiveness of an adapted form of the Center for the Promotion of Health in the New England Workplace (CPH-NEW) Healthy Workplace Participatory Program (HWPP) for strengthening cohesiveness, engagement, and impact of pre-existing joint labor-management health and safety committees.

The sites are enrolled in three pairs, matched by agency and type of services. For each pair of sites, one will be randomly selected for immediate HWPP coaching. The paired organization will serve as a control until the study mid-point, at which time all sites will be coached. Process evaluations will examine barriers to and facilitators of program uptake, reach, and effectiveness. Survey data and injury records will be examined in intervention and control groups to describe the frequencies of workplace and non-occupational exposures of selected health outcomes.

DETAILED DESCRIPTION:
Safety & Health through Integrated, Facilitated Teams (SHIFT) is a five-year study with etiologic, intervention, and translational research components. Six public sector healthcare institutions are enrolled, in three pairs matched by agency and type of services. The sites are four Massachusetts state healthcare facilities, which have recently been mandated by law to achieve "Occupational Health and Safety Administration (OSHA) equivalent compliance," and two Veterans Administration facilities each of which has multiple nationally mandated programs addressing employee health and safety. Using a "stepped wedge" design, one of each pair will be randomly selected as the immediate intervention site, while the other facility will be the concurrent control or "lagged intervention" site, having access only to technical reports and information until mid-project, when it will also receive the full intervention.

The intervention is the CPH-NEW Healthy Workplace Participatory Program (HWPP), a process for increasing the effectiveness of occupational health and safety committees or peer-led employee teams, through root cause analysis, prioritizing health and safety needs for effective problem-solving, identifying feasible interventions, and presenting these to leadership. Each facility has a pre-existing labor-management health and safety committee (HSC), which is the unit of intervention, so the HWPP will be adapted to joint management-labor teams. The committee is a partner in designing the program to fit the constraints and needs of the specific workplace and workforce. The research team provides training, coaching in the HWPP process, technical information, and practical assistance to committee members, facilitators, champions and leadership.

Etiologic research will entail analysis of baseline data for cross-sectional associations of work organization with worker health indicators. Intervention research will entail effectiveness and cost-outcome analysis of the HWPP. Outcomes will be both generic indicators of employee well-being and specific outcomes appropriate to the topics that the HSC's select for intervention. Translational research (process evaluation) will evaluate the efficacy of the dissemination and training strategy, as well as obstacles to and facilitators of uptake and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Direct employee of the agency (not temporary agency or subcontractor)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Team Attendance | Through study completion, an average of three years
  Attendance for each Design Team meeting (1-2 times per month)
Change in Team Engagement | Through study completion, an average of three years
  Percentage of yes responses for 2 survey items collected following Design Team meetings (1-2 times per month): "I spoke up and gave my opinion at this meeting" and "My opinion was considered seriously by others at this meeting." (Yes, no, somewhat). Items are computed individually.
Change in Level of Committee Activity | Through study completion, an average of three years
  A qualitative summary of field notes collected by research personnel following Design Team meetings (1-2 times per month) over the course of the study
Change in team-selected health/safety/well-being issue | Through study completion, an average of two years
  Targeted pre- and post-intervention surveys will be designed and administered by the Design Team

SECONDARY OUTCOMES:
Proportion of content followed according to the HWPP protocol | Through study completion, an average of three years
  A process measure that will be determined by adherence to HWPP protocol and pre-designed agendas for Design Team meetings (1-2 times per month)
Change in scope of health/safety/well-being | Through study completion, an average of three years
  Periodic interviews, designed by the research team, will be conducted with Design Team co-facilitators and Steering Committee Champions, and compared to results from baseline leadership interviews, designed by the research team, regarding scope of health/safety/well-being
Shared labor-management awareness of job-related health issues | Through study completion, an average of two years
  Interim interviews, designed by the research team, will be conducted with Design Team co-facilitators and Steering Committee Champions.
Work Ability of Employees | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes items from the Work Ability Index (Ilmarinen, 1991). Scores range from 7-49. Higher scores indicate better work ability.
Quality of Care of Patients/Residents: All-Employee Survey | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes three items related to quality of care from Aiken et al., 2002. Items are computed individually.
Organizational Support for Health, Safety, and Wellbeing | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes eight selected items from the Nordic Occupational Safety Climate Questionnaire (NOSACQ50). The score is an average of the 8 items. The score ranges from 1-4, where higher scores indicate better support from management for safety.
Employee Burnout: Exhaustion and Disengagement | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes 6 questions, 3 related to exhaustion and 3 related to disengagement (Demerouti, 2000; Halbeslebeni 2005). The score is an average of the items. The score ranges from 1-5, where higher scores indicate more exhaustion and more disengagement.
Frequency of Threats, Assault, and Harassment of Employees | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes 3 questions designed by the research team, including "In the past 6 months have you experienced someone who threatened to physically hurt or assault you?" "In the past 6 months have you experienced someone who did hurt or assault you?" "In the past 6 months have you experienced someone who sexually harassed you?" (Response categories: none, patient/family member/visitor, supervisor, other employee). Items are computed individually.
Change in Worker Injuries | Through study completion, an average of five years
  Annual rates of work-related injuries reported to the Workers' Compensation system - overall and by job type, and selected subgroups such as assault or back injury
Musculoskeletal Pain | Prior to random selection of immediate and delayed intervention site, and 3 years later
  The "All-Employee Survey" includes questions related to musculoskeletal pain in various body regions (low back, shoulder/upper arm, forearm/wrist/hand, knee, neck, ankle/foot) in the last three months. Level of discomfort (none, mild, moderate, severe, extreme) and measures of severity (use of pain relievers, surgery/physical therapy) are also included for each body region. Pain in each body region is computed individually.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Punnett, ScD, Principal Investigator — University of Massachusetts, Lowell

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Punnett L, Nobrega S, Zhang Y, Rice S, Gore R, Kurowski A; SHIFT Project Research Team. Safety and Health through Integrated, Facilitated Teams (SHIFT): stepped-wedge protocol for prospective, mixed-methods evaluation of the Healthy Workplace Participatory Program. BMC Public Health. 2020 Sep 29;20(1):1463. doi: 10.1186/s12889-020-09551-2. PMID 32993607